CLINICAL TRIAL: NCT02691702
Title: A Phase 1, Double Blind, Sponsor Open, Randomized, Placebo And Active Comparator Controlled, Dose Escalation Study To Investigate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Escalating Doses Of Pf-05251749 In Healthy Adult And Elderly Subjects
Brief Title: Multiple Dose Study Of BIIB118 (PF-05251749) In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B8001002; MAD (Other: Alias Study Number)
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Healthy Adult Subjects; Healthy Elderly Subjects
Keywords: Multiple Ascending Dose Study; Safety and Tolerability; Pharmacokinetics; Pharmacodynamics; Melatonin; Plasma; Dim Light Melatonin Onset
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Multiple Doses - Part A (Experimental): Multiple ascending doses administered in the morning to healthy adult subjects in a parallel study design
  Interventions: Drug: BIIB118; Drug: Melatonin
- Multiple Dose - Part B (Experimental): Multiple ascending doses administered in the evening to healthy adult subjects in a parallel study design
  Interventions: Drug: BIIB118
- Multiple Doses - Elderly (Experimental): Multiple ascending doses administered to elderly subjects
  Interventions: Drug: BIIB118

INTERVENTIONS:
Drug: BIIB118 — Multiple ascending doses of BIIB118 (50 mg, 150 mg, 450 mg and 900 mg) as extemporaneously prepared solution/suspension administered once daily over 2 weeks
  Other Names: PF-05251749
Drug: Melatonin — Positive control used to assess the validity of DLMO as pharmacodynamic endpoint.
  Arms: Multiple Doses - Part A

SUMMARY:
This is the first clinical trial to evaluate ascending multiple oral doses in healthy adult and healthy elderly subjects to characterize the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of BIIB118

DETAILED DESCRIPTION:
This study was previously posted by Pfizer. In March, 2020, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years (Parts A and B) or 65 and 85 years (Part C), inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Female subjects of non-childbearing potential must meet at least one of the following criteria:

  1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state;
  2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) will be considered to be of childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study medication (whichever is longer).
* Screening supine blood pressure >= 140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), repeat per local standard operating procedures (SOP). If orthostatic changes are present and deemed to be clinically significant by the investigator, Subject can be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - QPS-MRA, LLC (Miami Research Associates), South Miami, Florida
  - Qps-Mra, Llc, South Miami, Florida

REFERENCES:
- [Derived] Lin J, Gaudreault F, Johnson N, Lin Z, Nouri P, Goosen TC, Sawant-Basak A. Investigation of CYP3A induction by PF-05251749 in early clinical development: comparison of linear slope physiologically based pharmacokinetic prediction and biomarker response. Clin Transl Sci. 2022 Sep;15(9):2184-2194. doi: 10.1111/cts.13352. Epub 2022 Jul 2. PMID 35730131
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B8001002&StudyName=A+Phase+1%2C+Double+Blind%2C+Sponsor+Open%2C+Randomized%2C+Placebo+And+Active+Comparator+Controlled%2C+Dose+Escalation+Study+To+Investigate+The+Safety%2C+Tolerability%2C+Pharmacokinetics+And+Pharmacodynamics+Of+Multiple+Escalating+Doses+Of+Pf-05251749+In+Healthy+Adult+And+Elderly+Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Part A): Participants received placebo suspensions matched to PF-05251749 at 08:00 AM after an overnight fast on Days 1, 7, 14 (other doses were administered outside a window of ±2 hours of giving food), and also received placebo capsules matched to melatonin at 06:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- Melatonin 0.5 mg PM (Part A): Participants received placebo suspensions matched to PF-05251749 at 08:00 AM after an overnight fast on Days 1, 7, 14 (other doses were administered outside a window of ±2 hours of giving food), and also received melatonin 0.5 mg at 06:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- PF-05251749 50 mg AM (Part A): Participants received PF-05251749 50 mg orally at 08:00 AM after an overnight fast on Days 1, 7, 14 (other doses were administered outside a window of ±2 hours of giving food), and also received placebo capsules matched to melatonin at 06:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- PF-05251749 100 mg AM (Part A): Participants received PF-05251749 100 mg orally at 08:00 AM after an overnight fast on Days 1, 7, 14 (other doses were administered outside a window of ±2 hours of giving food), and also received placebo capsules matched to melatonin at 06:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- PF-05251749 200 mg AM (Part A): Participants received PF-05251749 200 mg orally at 08:00 AM after an overnight fast on Days 1, 7, 14 (other doses were administered outside a window of ±2 hours of giving food), and also received placebo capsules matched to melatonin at 06:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- PF-05251749 400 mg AM (Part A): Participants received PF-05251749 400 mg orally at 08:00 AM after an overnight fast on Days 1, 7, 14 (other doses were administered outside a window of ±2 hours of giving food), and also received placebo capsules matched to melatonin at 06:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- PF-05251749 750 mg AM (Part A): Participants received PF-05251749 750 mg orally at 08:00 AM after an overnight fast on Days 1, 7, 14 (other doses were administered outside a window of ±2 hours of giving food), and also received placebo capsules matched to melatonin at 06:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- Placebo (Part B): Participants received placebo suspensions matched to PF-05251749 at 6:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- PF-05251749 50 mg PM (Part B): Participants received PF-05251749 50 mg orally at 6:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- PF-05251749 200 mg PM (Part B): Participants received PF-05251749 200 mg orally at 6:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
- PF-05251749 500 mg PM (Part B): Participants received PF-05251749 500 mg orally at 6:00 PM outside a window of ±2 hours of giving food. Dosing continued every day until the final dose was administered on Day 14.
Period: Overall Study
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Started | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Completed | 8 | 10 | 7 | 8 | 8 | 5 | 5 | 12 | 6 | 6 | 6
Not Completed | 2 | 1 | 1 | 0 | 0 | 3 | 3 | 0 | 2 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B) | Total
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8 | 97
Age, Customized [Number; unit: participants]
  < 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 years | 6 | 7 | 1 | 5 | 0 | 3 | 4 | 7 | 3 | 6 | 4 | 46
  45-64 years | 4 | 4 | 7 | 3 | 8 | 5 | 4 | 5 | 5 | 2 | 4 | 51
  >= 65 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 5 | 1 | 3 | 2 | 1 | 0 | 2 | 15
  Male | 9 | 11 | 8 | 8 | 3 | 7 | 5 | 10 | 7 | 8 | 6 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 9 | 6 | 8 | 7 | 7 | 8 | 10 | 7 | 6 | 7 | 82
  Black | 3 | 2 | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Bond and Lader Visual Analogue Scale (BL-VAS) on Days 1, 4, 7, 10, 14, 15 and 16 - Alertness
Description: The Bond and Lader Visual Analogue Scales (VAS) monitored the subjective mood of each participant on 16 mood scales. Participants were asked to indicate on the VAS scale ranging from 0 to 100 mm about how they felt at the moment the scale was administered (example, alert/drowsy; calm/excited; content/tensed). The individual responses from the 16 mood scales were then combined to make three affective dimensions/subscales a) alertness (average of 9 items [total range 0 to 100, where each item is ordered so that higher scores indicated more alertness]), b) mood (average of 2 items [total range 0 to 100, where higher scores indicated elevated mood]), and c) calmness (average of 5 items [total range 0 to 100, where higher scores indicated more calmness]). Baseline is defined as the last available recording prior to dosing on Day 1.
Time Frame: Baseline (0h on Day 1), Day 1 (2h), Day 4 (1.5h), Day 7 (0h, 2h), Day 10 (1.5h), Day 14 (0h, 2h), Day 15 (0h) and Day 16 (0h).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Units on a scale
  Day 1 (2h): number analyzed (Participants) | 10 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
  Day 1 (2h) | 2.16 (7.405) | 7.50 (8.043) | 6.71 (12.314) | 3.50 (10.071) | 4.58 (9.472) | 4.05 (6.038) | 1.49 (11.514) | -0.08 (6.382) | -2.83 (7.314) | -6.04 (10.085) | -1.93 (7.953)
  Day 4 (1.5h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 6 | 12 | 8 | 6 | 8
  Day 4 (1.5h) | -0.61 (14.480) | 5.88 (8.943) | 6.46 (11.092) | 6.51 (11.209) | 3.48 (12.533) | 6.23 (8.043) | -14.45 (17.182) | -0.46 (7.105) | -0.25 (6.349) | 0.65 (8.135) | -3.00 (5.143)
  Day 7 (0h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 8 | 6 | 7
  Day 7 (0h) | -4.00 (22.474) | 3.76 (11.243) | 2.21 (12.305) | 6.96 (9.630) | 3.39 (12.541) | 6.54 (12.898) | -2.14 (9.437) | 1.23 (6.356) | -0.50 (6.514) | 0.23 (5.771) | -0.79 (5.109)
  Day 7 (2h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 8 | 6 | 7
  Day 7 (2h) | -2.87 (21.022) | -0.63 (20.162) | 4.03 (14.212) | 7.54 (9.519) | 2.76 (6.221) | 8.04 (11.784) | -10.92 (15.343) | 1.57 (5.817) | -1.25 (6.743) | -3.00 (11.517) | -4.93 (9.924)
  Day 10 (1.5h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 7 | 6 | 7
  Day 10 (1.5h) | -2.97 (20.833) | 4.76 (13.174) | 5.83 (12.879) | 6.20 (6.462) | 4.83 (7.288) | 7.51 (10.848) | -9.08 (21.071) | 1.31 (5.667) | -0.09 (7.507) | -0.82 (7.100) | -0.53 (6.265)
  Day 14 (0h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 14 (0h) | 1.19 (16.566) | 4.97 (10.320) | 5.68 (12.631) | 1.50 (5.458) | 2.96 (10.782) | 8.30 (11.045) | 5.12 (9.507) | 1.43 (5.532) | -1.93 (9.227) | 0.18 (10.212) | -0.89 (8.264)
  Day 14 (2h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 14 (2h) | -0.53 (17.945) | 7.18 (11.543) | 6.03 (13.385) | 1.75 (14.316) | 4.15 (11.839) | 6.16 (11.063) | 0.42 (5.971) | 2.83 (5.437) | 0.28 (3.998) | 2.25 (5.623) | -3.33 (8.503)
  Day 15 (0h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 15 (0h) | 1.55 (15.940) | 7.38 (10.892) | 3.51 (16.583) | 9.13 (10.092) | 2.13 (14.382) | 8.57 (12.525) | 9.20 (8.385) | 1.62 (5.057) | 1.07 (4.223) | 3.15 (3.971) | -1.93 (6.736)
  Day 16 (0h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 16 (0h) | 1.20 (17.347) | 10.64 (15.791) | 6.80 (15.431) | 9.04 (9.736) | 3.93 (11.931) | 8.39 (11.696) | 9.88 (8.410) | 1.33 (6.533) | 1.02 (3.170) | 8.37 (13.401) | 5.61 (6.812)

2. Primary Outcome: Change From Baseline for Bond and Lader Visual Analogue Scale (BL-VAS) on Days 1, 4, 7, 10, 14, 15 and 16 - Calmness
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Units on a scale
  Day 1 (2h): number analyzed (Participants) | 10 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
  Day 1 (2h) | 0.70 (7.997) | 1.45 (3.940) | 3.56 (16.668) | 13.88 (20.662) | 1.56 (1.522) | 2.25 (5.175) | 1.81 (9.509) | -0.38 (2.630) | -2.06 (6.032) | -15.31 (20.114) | -0.56 (3.774)
  Day 4 (1.5h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 6 | 12 | 8 | 6 | 8
  Day 4 (1.5h) | 1.00 (10.808) | 4.00 (12.092) | 7.50 (24.391) | 16.13 (22.448) | -1.75 (8.302) | 1.50 (1.732) | -11.25 (18.030) | 1.25 (8.081) | -1.75 (4.652) | -5.83 (10.405) | 1.19 (5.035)
  Day 7 (0h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 8 | 6 | 7
  Day 7 (0h) | -3.17 (20.352) | -3.85 (11.255) | 8.63 (24.013) | 13.44 (21.089) | 1.06 (2.129) | 0.50 (3.948) | -12.10 (25.289) | 1.08 (7.902) | -5.19 (14.258) | -4.00 (4.950) | 3.36 (10.351)
  Day 7 (2h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 8 | 6 | 7
  Day 7 (2h) | -2.22 (20.935) | 0.40 (10.572) | 7.56 (24.693) | 14.44 (20.859) | 1.44 (1.348) | 2.14 (2.593) | -13.30 (26.537) | 1.54 (8.349) | -2.31 (6.954) | -8.58 (9.881) | -1.21 (12.419)
  Day 10 (1.5h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 7 | 6 | 7
  Day 10 (1.5h) | -3.61 (19.816) | 0.75 (5.149) | 7.56 (24.943) | 13.75 (20.707) | 1.81 (1.751) | 1.71 (2.464) | -11.90 (27.220) | 2.46 (7.356) | -0.57 (6.194) | -5.33 (11.725) | 0.21 (16.820)
  Day 14 (0h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 14 (0h) | 0.88 (15.833) | 2.30 (8.629) | 6.88 (25.531) | 14.69 (21.457) | 1.94 (2.008) | -4.29 (14.502) | -10.30 (27.174) | 2.88 (7.227) | -2.58 (7.902) | -4.00 (9.391) | 2.86 (11.607)
  Day 14 (2h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 14 (2h) | 1.75 (12.961) | 2.00 (6.245) | 8.06 (24.282) | 15.25 (21.471) | 1.44 (2.178) | 2.71 (2.498) | -3.20 (8.213) | 3.54 (6.600) | -1.08 (4.042) | -4.75 (9.837) | 4.07 (9.467)
  Day 15 (0h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 15 (0h) | 2.19 (12.764) | 1.85 (8.564) | 9.63 (23.242) | 14.81 (21.032) | -3.25 (16.160) | 2.50 (3.594) | 6.80 (12.065) | 2.79 (7.402) | 0.17 (3.502) | 0.58 (3.456) | 4.86 (10.327)
  Day 16 (0h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 16 (0h) | 1.81 (14.609) | 0.30 (11.622) | 8.94 (23.542) | 16.13 (21.922) | 2.00 (1.927) | 2.21 (2.706) | 0.90 (21.927) | 2.88 (7.441) | -0.08 (2.957) | 2.67 (9.548) | 6.93 (11.745)

3. Primary Outcome: Change From Baseline for Bond and Lader Visual Analogue Scale (BL-VAS) on Days 1, 4, 7, 10, 14, 15 and 16- Mood
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Units on a scale
  Day 1 (2h): number analyzed (Participants) | 10 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
  Day 1 (2h) | 1.16 (4.480) | 5.16 (15.927) | 2.20 (12.642) | 2.03 (5.579) | 5.55 (13.357) | 3.25 (7.391) | 0.50 (8.384) | 0.32 (5.402) | -1.43 (5.432) | -7.80 (11.921) | -2.85 (10.557)
  Day 4 (1.5h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 6 | 12 | 8 | 6 | 8
  Day 4 (1.5h) | -1.42 (13.299) | 2.78 (15.744) | 1.85 (11.244) | 2.30 (12.752) | 6.84 (12.834) | 5.23 (7.530) | -12.73 (13.168) | 1.25 (5.218) | -3.13 (8.269) | -8.60 (12.057) | -1.73 (3.798)
  Day 7 (0h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 8 | 6 | 7
  Day 7 (0h) | -3.73 (17.841) | -1.86 (12.644) | 0.93 (12.440) | 6.20 (9.953) | 7.30 (13.407) | 5.83 (10.032) | -6.68 (11.595) | -0.45 (7.295) | -0.38 (4.313) | -4.90 (6.395) | -3.06 (3.878)
  Day 7 (2h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 8 | 6 | 7
  Day 7 (2h) | -3.00 (17.138) | 3.30 (14.328) | 6.65 (11.230) | 3.83 (8.980) | 6.30 (8.661) | 5.83 (9.082) | -10.84 (11.344) | 1.32 (5.811) | -2.83 (7.719) | -2.87 (3.110) | -10.00 (16.401)
  Day 10 (1.5h): number analyzed (Participants) | 9 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 7 | 6 | 7
  Day 10 (1.5h) | -3.84 (18.444) | 2.12 (16.892) | 3.50 (11.745) | 5.13 (8.561) | 8.13 (12.784) | 6.11 (8.896) | -9.92 (17.802) | 1.50 (5.784) | -0.29 (4.783) | -3.97 (7.816) | -2.94 (1.672)
  Day 14 (0h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 14 (0h) | -3.65 (16.044) | 4.64 (14.753) | 5.13 (8.037) | 2.85 (8.854) | 6.33 (13.084) | 3.97 (11.878) | -0.84 (7.942) | 2.17 (6.178) | -2.20 (6.950) | -3.50 (8.772) | -2.09 (7.061)
  Day 14 (2h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 14 (2h) | -2.45 (19.691) | 5.54 (14.101) | 3.63 (12.086) | 6.88 (8.256) | 5.03 (14.154) | 4.46 (6.410) | -2.96 (4.883) | 2.10 (5.706) | -0.73 (3.259) | -2.03 (4.094) | -2.89 (6.350)
  Day 15 (0h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 15 (0h) | -1.15 (15.899) | 6.52 (14.121) | 4.70 (14.515) | 7.13 (9.288) | 3.25 (14.971) | 6.51 (9.306) | 2.80 (7.053) | 0.78 (7.989) | -0.30 (3.067) | 3.90 (10.749) | -1.26 (5.991)
  Day 16 (0h): number analyzed (Participants) | 8 | 10 | 8 | 8 | 8 | 7 | 5 | 12 | 6 | 6 | 7
  Day 16 (0h) | -1.38 (17.722) | 7.48 (19.847) | 7.36 (12.735) | 10.70 (6.978) | 4.95 (15.441) | 3.63 (6.738) | 3.00 (5.829) | 0.93 (7.767) | -0.20 (2.154) | 6.60 (17.980) | 1.74 (5.754)

4. Primary Outcome: Number of Participants With New Onset and Worsening of Post-baseline Suicidality for Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS was an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced any of the following 1: completed suicide, 2: suicide attempt (response of "yes" on "actual attempt"), 3: preparatory acts toward imminent suicidal behavior ("yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior"), 4: any suicidal behavior or ideation, suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent"), 7: self-injurious behavior, no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior"). The new onset and worsening of post-baseline suicidality for C-SSRS was reported.
Time Frame: Days 0, 7, 14, 16, and follow-up visit (28 calender days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants
  Day 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) (All Causalities)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage.
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants | 4 | 3 | 3 | 1 | 5 | 7 | 7 | 3 | 5 | 2 | 8

6. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) (Treatment Related)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; The event has a causal relationship with the treatment or usage.
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants | 1 | 2 | 2 | 1 | 1 | 5 | 7 | 2 | 4 | 2 | 8

7. Primary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: The laboratory test included: hematology (hemoglobin, hematocrit, red blood cell count, MCV, MCH, MCHC, platelets, white blood cell count, absolute lymphocytes, absolute total neutrophils, absolute basophils, absolute eosinophils and absolute monocytes), coagulation (PPT, prothrombin, PT international, ratio and fibrinogen, liver function(total bilirubin, direct bilirubin, aspartate, AST, Alanine, ALT, gamma GT, alkaline phosphatase, total protein and albumin), renal function (blood urea nitrogen, creatinine, HDL cholesterol, LDL cholesterol, triglycerides), Electrolytes (sodium, potassium, chloride, calcium, phosphate, venous bicarbonate), clinical chemistry (glucose, creatinine kinase), urinalysis dipstick (urine PH, urine glucose, urine ketones, urine protein, urine blood, urine urobilinogen, urine nitrite, urine leukocyte, esterase), urinalysis microscopy (urine RBC, urine WBC, urine casts, urine bacteria), miscellaneous (absolute lymphocyte marker CD4, CD8, CD19)
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants | 2 | 8 | 1 | 2 | 4 | 4 | 7 | 8 | 5 | 5 | 7

8. Primary Outcome: Number of Participants With Vital Signs Data Meeting Categorical Criteria (Absolute Values)
Description: Number of participants with vital signs data of absolute values meeting categorical criteria was reported as following: (1) Supine systolic BP < 90 mmHg; (2) Supine Diastolic BP < 50 mmHg; (3) Supine Pulse Rate < 40 BPM ; (4) Supine Pulse Rate > 120 BPM.
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants
  Supine Systolic BP < 90 mmHg | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Supine Diastolic BP < 50 mmHg | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Supine Pulse Rate < 40 BPM | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Pulse Rate > 120 BPM | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

9. Primary Outcome: Number of Participants With Vital Signs Data Meeting Categorical Criteria (Increases From Baseline)
Description: Number of participants with vital signs data of increase from baseline meeting the following criteria was reported: Criterion A: maximum increase from baseline in supine systolic BP >= 30 mmHg; Criterion B: maximum increase from baseline in supine diastolic BP >= 20 mmHg. Baseline was defined as the last available recording prior to dosing.
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants
  Criterion A | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Criterion B | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Vital Signs Data Meeting Categorical Criteria (Decrease From Baseline)
Description: Number of participants with vital signs data of increase from baseline meeting the following criteria was reported: Criterion A: maximum decrease from baseline in supine systolic BP >= 30 mmHg; Criterion B: maximum decrease from baseline in supine diastolic BP >= 20 mmHg. Baseline was defined as the last available recording prior to dosing.
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants
  Criterion A | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1
  Criterion B | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Categorical Criteria (Absolute Values)
Description: Number of participants with ECG data of absolute values meeting categorical criteria was reported as following: Criterion A: maximum PR interval (time from the beginning of P wave to the start of QRS complex, corresponding to the end of atrial depolarization and onset of ventricular depolarization) >= 300 msec; Criterion B: maximum QRS complex (time from Q wave to the end of S wave, corresponding to ventricle depolarization)>= 140 msec; Criterion C: Maximum QT interval (time from the beginning of Q wave to the end of T wave corresponding to electrical systole)>= 500 msec; Criterion D: maximum QTC interval (QT interval corrected for heart rate) 450-<480 msec; Criterion E: maximum QTC interval 480-<500 msec; Criterion F: maximum QTC interval >=500 msec; Criterion G: maximum QTCF interval (QT interval corrected for heart rate using Fridericia's formula) 450 -< 480 msec; Criterion H: maximum QTCF interval 480 -< 500 msec; Criterion I: maximum QTCF interval >=500 msec.
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants
  Criterion A | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion B | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion C | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion D | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Criterion E | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion F | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion G | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Criterion H | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion I | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Categorical Criteria (Increase From Baseline)
Description: Number of participants with ECG Data of increase from baseline meeting the following criteria was reported: Criterion A: maximum PR interval increase from baseline percentage change (PctChg)>=25/50%; Criterion B: maximum QRS complex increase from baseline PctChg >=50%; Criterion C: maximum QTC interval (time from the beginning of Q wave to the end of T wave corresponding to electrical systole, corrected for heart rate) increase from baseline 30<=change<60 msec; Criterion D: maximum QTC interval increase from baseline change >=60 msec; Criterion E: maximum QTCF (Fridericia's correction) interval increase from baseline 30<=change<60; Criterion F: maximum QTCF interval increase from baseline change >=60 msec. Baseline was defined as the average of the triplicate measurements prior to dosing on Day 1.
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants
  Criterion A | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion B | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion C | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 0
  Criterion D | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion E | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 0
  Criterion F | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With New/Intensified Physical Examination Findings
Description: Physical examination included examination of ears, eyes, gastrointestinal, head, heart, lungs, lymph nodes, mouth, musculoskeletal, nose, skin. The number of participants with new-intensified physical examination findings were reported.
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With New/Intensified Neurological Examination Findings
Description: The number of participants with new-intensified neurological examination findings were reported.
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Population: The safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 10 | 11 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-05251749 - Days 1, 7 and 14
Description: Maximum plasma concentration (Cmax) of PF-05251749 was observed directly from data on Days 1, 7 and 14.
Time Frame: Days 1 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 48h), 7 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24h) and 14 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 48h).
Population: The Pharmacokinetic (PK) concentration population was defined as all enrolled participants treated who received at least 1 dose of PF-05251749 and had at least 1 measureable concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/mililiter (ng/mL)
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
nanogram/mililiter (ng/mL)
  Day 1 | 346.1 (36) | 838.1 (29) | 1600 (33) | 2465 (36) | 3990 (17) | 219.4 (23) | 898.0 (23) | 1833 (44)
  Day 7: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 7
  Day 7 | 440.6 (23) | 971.6 (26) | 1583 (24) | 2917 (36) | 4428 (22) | 239.3 (19) | 1018 (29) | 2747 (42)
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 6 | 6 | 7
  Day 14 | 420.9 (42) | 1068 (25) | 1907 (17) | 2613 (28) | 4726 (19) | 271.0 (22) | 904.3 (55) | 2714 (60)

16. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to Tau (AUCtau) of PF-05251749 - Days 1, 7 and 14.
Description: AUCtau referred to the area under the curve from time 0 to time tau, the dosing interval, where tau equaled to 24 hours on Days 1, 7 and 14.
Time Frame: as for outcome 15
Population: The PK parameter population was defined as all enrolled participants treated who received at least 1 dose of PF-05251749 and had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/mililiter (ng*hr/mL)
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
nanogram*hour/mililiter (ng*hr/mL)
  Day 1 | 1430 (39) | 3302 (29) | 6514 (21) | 14060 (31) | 26630 (25) | 1626 (27) | 6385 (29) | 16210 (31)
  Day 7: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 7 | 6 | 7
  Day 7 | 1700 (31) | 4260 (20) | 7662 (25) | 15970 (31) | 32890 (34) | 1801 (21) | 7018 (28) | 18720 (37)
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 6 | 6 | 7
  Day 14 | 1619 (37) | 4234 (19) | 8503 (24) | 13640 (28) | 33290 (17) | 1869 (24) | 6778 (35) | 21950 (50)

17. Secondary Outcome: Time at Which Cmax Occurred (Tmax) of PF-05251749 - Days 1, 7 and 14
Description: Tmax of PF-05251749 was observed directly from data on Days 1, 7 and 14, as time of first occurrence.
Time Frame: as for outcome 15
Population: as for outcome 16
Measure: Median (Full Range); unit: hr
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
hr
  Day 1 | 1.00 [0.500 to 1.00] | 1.00 [0.500 to 1.50] | 1.00 [0.500 to 1.00] | 1.00 [1.00 to 3.00] | 1.00 [0.500 to 3.00] | 1.75 [1.00 to 3.00] | 1.00 [0.500 to 3.00] | 1.00 [0.500 to 12.0]
  Day 7: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 7
  Day 7 | 0.500 [0.500 to 2.00] | 1.00 [0.500 to 1.50] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 3.00] | 1.50 [1.00 to 3.00] | 1.00 [1.00 to 3.00] | 0.750 [0.450 to 3.00] | 1.50 [0.500 to 3.00]
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 6 | 6 | 7
  Day 14 | 1.00 [0.500 to 1.00] | 1.00 [0.500 to 1.00] | 1.00 [0.500 to 1.50] | 1.00 [0.500 to 2.00] | 1.00 [0.500 to 1.00] | 1.00 [0.500 to 1.50] | 2.00 [0.500 to 3.00] | 2.00 [1.00 to 3.00]

18. Secondary Outcome: Apparent Clearance (CL/F) of PF-05251749 - Days 7 and 14
Description: Apparent clearance was influenced by the fraction of the dose absorbed, which was measured by Dose/AUCtau.
Time Frame: Days 7 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24h) and 14 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 48h).
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/hr)
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Liter/hour (L/hr)
  Day 7: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 7 | 6 | 7
  Day 7 | 29.42 (31) | 23.49 (20) | 26.09 (25) | 25.08 (31) | 22.76 (34) | 27.76 (21) | 28.50 (28) | 26.74 (38)
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 6 | 6 | 7
  Day 14 | 30.86 (37) | 23.61 (19) | 23.53 (24) | 29.34 (28) | 22.51 (17) | 26.76 (23) | 29.54 (34) | 22.82 (51)

19. Secondary Outcome: Minimum Concentration Observed (Cmin) of PF-05251749 - Days 7 and 14
Description: Minimum concentration observed (Cmin) of PF-05251749 was observed directly from data on Days 7 and 14.
Time Frame: Days 7 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24h) and 14 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 48h).
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng/mL
  Day 7: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 7
  Day 7 | 11.01 (49) | 27.35 (41) | 65.88 (46) | 114.9 (75) | 340.3 (99) | 19.48 (24) | 53.88 (26) | 161.6 (100)
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 6 | 6 | 7
  Day 14 | 11.40 (51) | 28.89 (38) | 79.56 (46) | 96.98 (64) | 375.7 (59) | 19.11 (45) | 56.77 (24) | 178.6 (105)

20. Secondary Outcome: Plasma Peak-to-trough Ratio (PTR) (Cmax/Cmin) of PF-05251749 - Days 7 and 14
Description: Peak-to-through ratio (PTR) was the ratio of Cmax to Cmin, which was measured on Days 7 and 14.
Time Frame: Days 7 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24h) and 14 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 48h).
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Ratio
  Day 7: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 7
  Day 7 | 40.04 (41) | 35.54 (51) | 24.01 (39) | 25.37 (72) | 13.00 (81) | 12.29 (19) | 18.90 (24) | 17.02 (63)
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 6 | 6 | 7
  Day 14 | 36.93 (18) | 36.98 (33) | 23.98 (35) | 26.92 (65) | 12.57 (64) | 14.17 (49) | 15.92 (34) | 15.20 (101)

21. Secondary Outcome: Observed Accumulation Ratio (Rac) of PF-05251749 -Days 7 and 14
Description: Observed accumulation ratio (Rac) was calculated as AUCtau (Days 7 or 14) divided by AUCtau (Day 1).
Time Frame: Days 7 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24h) and 14 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 48h).
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Ratio
  Day 7: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 7 | 6 | 7
  Day 7 | 1.188 (16) | 1.289 (13) | 1.176 (9) | 1.160 (17) | 1.255 (7) | 1.169 (12) | 1.097 (7) | 1.205 (14)
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 6 | 6 | 7
  Day 14 | 1.133 (17) | 1.283 (19) | 1.307 (15) | 0.9892 (16) | 1.270 (21) | 1.195 (12) | 1.061 (9) | 1.414 (20)

22. Secondary Outcome: Observed Accumulation Ratio for Cmax (Rac,Cmax) of PF-05251749 - Days 7 and 14
Description: Observed accumulation ratio for Cmax (Rac,Cmax) was calculated as: Cmax on Day 7 or 14 divided by Cmax on Day 1.
Time Frame: Days 7 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24h) and 14 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 48h).
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Ratio
  Day 7: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 7
  Day 7 | 1.272 (27) | 1.160 (14) | 0.9898 (21) | 1.161 (34) | 1.155 (10) | 1.093 (12) | 1.090 (28) | 1.422 (52)
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 6 | 6 | 7
  Day 14 | 1.216 (35) | 1.273 (28) | 1.194 (27) | 1.039 (20) | 1.234 (19) | 1.226 (13) | 0.9686 (47) | 1.404 (21)

23. Secondary Outcome: Terminal Half-Life (t1/2) of PF-05251749 - Day 14
Description: Terminal half-life (t1/2) was calculated as Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: Day 14 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 48h).
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
hr | 9.625 (2.0701) | 9.630 (1.6523) | 10.91 (1.4405) | 9.940 (2.3215) | 11.20 (3.0942) | 10.62 (1.4922) | 8.878 (0.93101) | 10.62 (2.1519)

24. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-05251749 - Day 14
Description: Apparent volume of distribution (Vz/F) was calculated by Dose/(AUCtau × kel) on Day 14.
Time Frame: Day 14 (0, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 48h).
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
L | 419.3 (39) | 323.6 (27) | 363.9 (21) | 409.0 (43) | 353.6 (17) | 405.5 (14) | 376.5 (42) | 343.9 (36)

25. Secondary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine Over Dosing Interval Tau (Aetau) of PF-05251749 - Day 14
Description: Aetau was the cumulative amount of drug recovered unchanged in urine from time 0 to end of the dosing interval, which was calculated by sum of (urine concentration × volume of urine).
Time Frame: Day 14 (0, 0.5, 1, 1.5, 2, 3, 4, 5, 8, 12, 16, 20, 24, 48h).
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
ng | 56710 (39) | 142900 (31) | 317900 (41) | 404900 (59) | 738300 (40)

26. Secondary Outcome: Percentage of Dose Recovered Unchanged in Urine Over Dosing Interval Tau (Aetau%) of PF-05251749 - Day 14
Description: Aetau% was the percentage of dose recovered unchanged into urine from 0 to end of the dosing interval, which was calculated by 100 × Aetau/Dose.
Time Frame: Day 14 (0, 0.5, 1, 1.5, 2, 3, 4, 5, 8, 12, 16, 20, 24, 48h).
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of PF-05251749
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Percentage of PF-05251749 | 0.1133 (39) | 0.1429 (31) | 0.1591 (41) | 0.1013 (59) | 0.09849 (41)

27. Secondary Outcome: Renal Clearance (CLr) of PF-05251749 - Day 14
Description: Renal clearance was calculated as cumulative amount of drug recovered unchanged in urine during the dosing interval (Ae) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCtau), Aetau/AUCtau.
Time Frame: Day 14 (0, 0.5, 1, 1.5, 2, 3, 4, 5, 8, 12, 16, 20, 24, 48h).
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
mL/hr | 37.18 (44) | 33.76 (33) | 37.39 (36) | 29.73 (30) | 22.15 (31)

28. Secondary Outcome: Change From Baseline for Dim Light Melatonin Onset (DLMO) Time - Day 6
Description: Dim Light Melatonin Onset (DLMO) was defined as point in time when the smooth melatonin curve exceeds the threshold. The threshold for each melatonin profile was calculated as the mean of three low consecutive daytime values (raw data points) plus twice the standard deviation of these points.
Time Frame: Day 0 (Baseline) and Day 6.
Population: The PD (pharmacodynamic) population was defined as all enrolled participants treated who provided at least 3 measurable salivary melatonin concentrations.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 9 | 10 | 8 | 6 | 8 | 8 | 7 | 12 | 8 | 8 | 8
min | 10.0 (45.17) | 3.3 (64.42) | 11.3 (45.18) | 37.5 (78.90) | 85.0 (83.61) | 124.3 (61.06) | 150.0 (56.12) | 13.6 (64.85) | 86.3 (84.00) | 135.0 (88.49) | 205.0 (44.16)
Statistical Analysis 1: Comparison: Placebo (Part A) vs Melatonin 0.5 mg PM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = -1.26, 90% CI 2-sided [-63.09 to 60.57], Standard Error of Mean 37.24 — Test (Melatonin 0.5 mg PM) Reference (Placebo)
Statistical Analysis 2: Comparison: Placebo (Part A) vs PF-05251749 50 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = -27.13, 90% CI 2-sided [-91.24 to 36.97], Standard Error of Mean 38.61 — Test (PF-05251749 50 mg AM) Reference (Placebo)
Statistical Analysis 3: Comparison: Placebo (Part A) vs PF-05251749 100 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = 43.72, 90% CI 2-sided [-32.19 to 119.62], Standard Error of Mean 45.72 — Test (PF-05251749 100 mg AM) Reference (Placebo)
Statistical Analysis 4: Comparison: Placebo (Part A) vs PF-05251749 200 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = 61.48, 90% CI 2-sided [-6.38 to 129.35], Standard Error of Mean 40.88 — Test (PF-05251749 200 mg AM) Reference (Placebo)
Statistical Analysis 5: Comparison: Placebo (Part A) vs PF-05251749 400 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = 125.87, 90% CI 2-sided [60.51 to 191.23], Standard Error of Mean 39.37 — Test (PF-05251749 400 mg AM) Reference (Placebo)
Statistical Analysis 6: Comparison: Placebo (Part A) vs PF-05251749 750 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = 156.22, 90% CI 2-sided [84.99 to 227.45], Standard Error of Mean 42.91 — Test (PF-05251749 750 mg AM) Reference (Placebo)
Statistical Analysis 7: Comparison: Placebo (Part B) vs PF-05251749 50 mg PM (Part B); Test type: Other — MMRM; Mean Difference (Final Values) = 51.42, 90% CI 2-sided [-3.57 to 106.41], Standard Error of Mean 33.12 — Test (PF-05251749 50 mg PM) Reference (Placebo)
Statistical Analysis 8: Comparison: Placebo (Part B) vs PF-05251749 200 mg PM (Part B); Test type: Other — MMRM; Mean Difference (Final Values) = 142.74, 90% CI 2-sided [82.76 to 202.72], Standard Error of Mean 36.13 — Test (PF-05251749 200 mg PM) Reference (Placebo)
Statistical Analysis 9: Comparison: Placebo (Part B) vs PF-05251749 500 mg PM (Part B); Test type: Other — MMRM; Mean Difference (Final Values) = 174.90, 90% CI 2-sided [115.11 to 234.69], Standard Error of Mean 36.01 — Test (PF-05251749 500 mg PM) Reference (Placebo)

29. Secondary Outcome: Change From Baseline for Dim Light Melatonin Onset (DLMO) Time - Day 15
Description: DLMO was defined as point in time when the smooth melatonin curve exceeds the threshold. The threshold for each melatonin profile was calculated as the mean of three low consecutive daytime values (raw data points) plus twice the standard deviation of these points.
Time Frame: Day 0 (Baseline) and Day 15
Population: The PD population was defined as all enrolled participants treated who provided at least 3 measurable salivary melatonin concentrations.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
Number analyzed (Participants) | 9 | 10 | 8 | 6 | 8 | 8 | 7 | 12 | 8 | 8 | 8
min | 40.0 (61.97) | -36.7 (93.41) | 56.3 (54.23) | 112.5 (75.00) | 100.0 (137.70) | 115.7 (118.02) | 150.0 (56.12) | 49.1 (103.29) | 150.0 (73.48) | 135.0 (88.49) | 210.0 (47.43)
Statistical Analysis 1: Comparison: Placebo (Part A) vs Melatonin 0.5 mg PM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = -71.26, 90% CI 2-sided [-133.09 to -9.43], Standard Error of Mean 37.24 — Test (Melatonin 0.5 mg PM) Reference (Placebo)
Statistical Analysis 2: Comparison: Placebo (Part A) vs PF-05251749 50 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = -12.13, 90% CI 2-sided [-76.24 to 51.97], Standard Error of Mean 38.61 — Test (PF-05251749 50 mg AM) Reference (Placebo)
Statistical Analysis 3: Comparison: Placebo (Part A) vs PF-05251749 100 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = 88.72, 90% CI 2-sided [12.81 to 164.62], Standard Error of Mean 45.72 — Test (PF-05251749 100 mg AM) Reference (Placebo)
Statistical Analysis 4: Comparison: Placebo (Part A) vs PF-05251749 200 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = 46.48, 90% CI 2-sided [-21.38 to 114.35], Standard Error of Mean 40.88 — Test (PF-05251749 200 mg AM) Reference (Placebo)
Statistical Analysis 5: Comparison: Placebo (Part A) vs PF-05251749 400 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = 87.30, 90% CI 2-sided [21.94 to 152.66], Standard Error of Mean 39.37 — Test (PF-05251749 400 mg AM) Reference (Placebo)
Statistical Analysis 6: Comparison: Placebo (Part A) vs PF-05251749 750 mg AM (Part A); Test type: Other — MMRM; Mean Difference (Final Values) = 126.22, 90% CI 2-sided [54.99 to 197.45], Standard Error of Mean 42.91 — Test (PF-05251749 750 mg AM) Reference (Placebo)
Statistical Analysis 7: Comparison: Placebo (Part B) vs PF-05251749 50 mg PM (Part B); Test type: Other — MMRM; Mean Difference (Final Values) = 92.36, 90% CI 2-sided [33.51 to 151.21], Standard Error of Mean 35.48 — Test (PF-05251749 50 mg PM) Reference (Placebo)
Statistical Analysis 8: Comparison: Placebo (Part B) vs PF-05251749 200 mg PM (Part B); Test type: Other — MMRM; Mean Difference (Final Values) = 107.29, 90% CI 2-sided [47.31 to 167.27], Standard Error of Mean 36.13 — Test (PF-05251749 200 mg AM) Reference (Placebo)
Statistical Analysis 9: Comparison: Placebo (Part B) vs PF-05251749 500 mg PM (Part B); Test type: Other — MMRM; Mean Difference (Final Values) = 140.61, 90% CI 2-sided [77.91 to 203.30], Standard Error of Mean 37.79 — Test (PF-05251749 500 mg AM) Reference (Placebo)

ADVERSE EVENTS:
Time Frame: Day 1 to follow-up visit (28 calendar days after the last dose of investigational product on Day 14).
Arm/Group | Placebo (Part A) | Melatonin 0.5 mg PM (Part A) | PF-05251749 50 mg AM (Part A) | PF-05251749 100 mg AM (Part A) | PF-05251749 200 mg AM (Part A) | PF-05251749 400 mg AM (Part A) | PF-05251749 750 mg AM (Part A) | Placebo (Part B) | PF-05251749 50 mg PM (Part B) | PF-05251749 200 mg PM (Part B) | PF-05251749 500 mg PM (Part B)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 1/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/10 | 3/11 | 3/8 | 1/8 | 5/8 | 7/8 | 7/8 | 3/12 | 4/8 | 2/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A) (N=10) | Melatonin 0.5 mg PM (Part A) (N=11) | PF-05251749 50 mg AM (Part A) (N=8) | PF-05251749 100 mg AM (Part A) (N=8) | PF-05251749 200 mg AM (Part A) (N=8) | PF-05251749 400 mg AM (Part A) (N=8) | PF-05251749 750 mg AM (Part A) (N=8) | Placebo (Part B) (N=12) | PF-05251749 50 mg PM (Part B) (N=8) | PF-05251749 200 mg PM (Part B) (N=8) | PF-05251749 500 mg PM (Part B) (N=8)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A) (N=10) | Melatonin 0.5 mg PM (Part A) (N=11) | PF-05251749 50 mg AM (Part A) (N=8) | PF-05251749 100 mg AM (Part A) (N=8) | PF-05251749 200 mg AM (Part A) (N=8) | PF-05251749 400 mg AM (Part A) (N=8) | PF-05251749 750 mg AM (Part A) (N=8) | Placebo (Part B) (N=12) | PF-05251749 50 mg PM (Part B) (N=8) | PF-05251749 200 mg PM (Part B) (N=8) | PF-05251749 500 mg PM (Part B) (N=8)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 0 | 4
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
From Parts A and B, it was deemed that safety, tolerability, PK and PD objectives were met, so Part C was not conducted. Because of limited saliva sampling duration (06:00 PM to 12:00 AM), DLMO observation(s) beyond midnight could not be quantified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.